CLINICAL TRIAL: NCT02193789
Title: The Effect of Newly Designed Covered Self-expandable Metallic Stents Insertion Using Clips and Suture Materials for Preventing Migration in Benign Stricture of Gastroduodenal Anastomosis: a Pilot Study
Brief Title: Covered Self-expandable Metallic Stents Insertion Using Clips and Suture Materials for Preventing Migration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Kee Myung Lee, Professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-MDB-14-059
Record Dates: First submitted 2014-07-01; First posted 2014-07-18 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Gastroduodenal Anastomosis
Keywords: Anastomosis site structure; Stent insertion; Stent migration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anastomosis site stricture (Experimental): anastomosis site stricture after subtotal gastrectomy with Billroth-I anastomosis
  Interventions: Procedure: deployment of through the scope covered metallic stent at the stricture site; Device: Covered Self-expandable Metallic Stents

INTERVENTIONS:
Procedure: deployment of through the scope covered metallic stent at the stricture site — Deployment of Covered Self-expandable Metallic Stents Insertion fixing with Clips and Suture Material at the stricture site
Device: Covered Self-expandable Metallic Stents

SUMMARY:
In patients of subtotal gastrectomy with Billroth-I or Billroth-II anastomosis, Anastomosis site stricture is very severe complication. It can improve by temporary through the scope covered metallic stent. It is very effective procedure about the stricture. But stent migration is very severe complication. Herein the investigators suggest newly method to prevent the stent migration. Fixation of stent by hemoclip is effective method to prevent stent migration. But it is difficult to remove stent after resolved stricture. So the investigators add the suture between hemoclip and stent. And the investigators cut the suture when stent removal.

ELIGIBILITY:
Inclusion Criteria:

* subtotal gastrectomy with Billroth-I or Billroth-II anastomosis
* symptom of gastric outlet obstruction
* anastomosis site stricture after surgery

Exclusion Criteria:

* patients of the impossible stent insertion due to other complication
* foreigner
* no agree a concent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Improvement of symptom (Resolving anastomosis site stricture) | Up to 1 month
  Improvement of food intake. It was measured by the gastric outlet obstruction scoring system (GOOSS) score, with 0 = no oral intake, 1 = liquid diet, 2 = soft diet, and 3 = regular diet.

SECONDARY OUTCOMES:
Complications associated with the procedure | Up to 1 month (time of stent removal)
  Check all the complications associated with the procedure (e.g. procedure failure, stent migration, no improvement of symptom, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Gyo Lim, M.D., Principal Investigator — Ajou University School of Medicine; Ki Seong Lee, M.D., Principal Investigator — Ajou University School of Medicine; Joon Koo Kang, M.D., Principal Investigator — Ajou University School of Medicine
Locations (2):
- South Korea (2):
  - Ajou university hospital, Suwon, Gyeong-gi Do
  - Ajou University Hospital, Suwon